CLINICAL TRIAL: NCT02004392
Title: A 26-Week Extension Study of the Safety and Clinical Effects of EVP-6124 in Subjects With Alzheimer's Disease Currently or Previously Receiving an Acetylcholinesterase Inhibitor Medication
Brief Title: Study of the Safety and Clinical Effects of 2 Doses of EVP-6124 in Subjects With Alzheimer's Disease Who Complete Study EVP-6124-024 or EVP-6124-025
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Study has been suspended due to clinical hold.
Sponsor: FORUM Pharmaceuticals Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: EVP-6124-026; 2013-002654-75 (EudraCT Number)
Record Dates: First submitted 2013-11-27; First posted 2013-12-09 (Estimated); Last update posted 2016-05-03 (Estimated); Status verified 2015-09

CONDITIONS: Alzheimer's Disease; Dementia
Keywords: Alzheimer's disease; Cognition; Alpha-7 nAChR
MeSH Terms: conditions — Alzheimer Disease; Dementia | interventions — 7-chloro-N-quinuclidin-3-yl-benzo(b)thiophene-2-carboxamide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EVP-6124, low dose (Experimental): low dose, Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: EVP-6124
- EVP-6124, high dose (Experimental): high dose, Tablet, Once Daily, Day 1 through Day 182
  Interventions: Drug: EVP-6124

INTERVENTIONS:
Drug: EVP-6124

SUMMARY:
This is a 26-week, randomized extension of the Phase 3 double-blind placebo-controlled studies, EVP-6124-024 and EVP-6124-025. In this extension study, subjects who complete study EVP-6124-024 or EVP-6124-025 and fulfill all entry criteria will be randomized to receive EVP-6124 for an additional 26 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects of any race, aged ≥55 and ≤85 years at time of entry into study EVP-6124-024 or EVP-6124-025
* Informed consent form (ICF) for this extension study signed by the subject or legally acceptable representative and an ICF signed by the support person/caregiver before initiation of any study-specific procedures
* Successful completion (Day 182) of study EVP-6124-024 or EVP-6124-025
* No clinically significant change in the judgment of the investigator in the subject's medical status during study EVP-6124-024 or EVP-6124-025
* In the judgment of the investigator, extension treatment is in the best interest of the subject
* Fertile, sexually active subjects (men and women) must use an effective method of contraception during the study. Female subjects and the female partner of male subjects must be surgically sterile (hysterectomy or bilateral tubal ligation), postmenopausal for at least 1-year, or willing to practice adequate methods of contraception if of childbearing potential (defined as consistent use of combined effective methods of contraception [including at least 1 barrier method])
* Reliable and capable support person/caregiver, who if not living in the same household, interacts with the subject approximately 4 times per week and will be available to attend clinic visits in person when possible

Exclusion Criteria:

* Significant risk of suicidal or violent behavior in the judgment of the investigator
* Adverse events from the previous study (EVP-6124-024 or EVP-6124-025) that have not resolved, are moderate or severe, judged to be possibly related or related to study drug, and considered by the investigator to be a contraindication to extension study participation
* Any condition that would make the subject in the judgment of the investigator unsuitable for the study
* Female subjects who are pregnant, nursing, or planning to become pregnant during the extension study

Ages: 55 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 348 (Actual)
Dates: Start 2014-06; Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Safety of 2 fixed doses of EVP-6124 for up to 52 weeks in subjects with Alzheimer's disease who complete study EVP-6124-024 or EVP-6124-025 | Baseline to Day 182 or Early Termination
  Criteria for evaluation include: adverse events, clinical laboratory tests, vital signs, body weight, 12-lead ECG, physical examination, concomitant medications, C-SSRS, and GDS.

SECONDARY OUTCOMES:
Change from Baseline in cognition using the Mini-Mental State Examination (MMSE) | Baseline to Day 182 or Early Termination
Change from Baseline in psychiatric and behavioral symptoms using the Neuropsychiatric Inventory (NPI) | Baseline to Day 182 or Early Termination
Change from Baseline in quality of life using the EuroQol-5D (EQ-5D) | Baseline to Day 182 or Early Termination
Pharmacoeconomic outcomes using the Resource Utilization in Dementia (RUD-Lite 3.3) | Baseline to Day 182 or Early Termination
Caregiver perceived burden using the Zarit Burden Interview (ZBI) | Baseline to Day 182 or Early Termination

CONTACTS AND LOCATIONS:
Locations (86):
- United States (56):
  - Phoenix, Arizona
  - Tucson, Arizona
  - Little Rock, Arkansas
  - Costa Mesa, California
  - Culver City, California
  - Encino, California
  - Glendale, California
  - Long Beach, California
  - Los Alamitos, California
  - Orange, California
  - Redding, California
  - San Diego, California
  - New Haven, Connecticut
  - Norwich, Connecticut
  - Atlantis, Florida
  - Brooksville, Florida
  - Delray Beach, Florida
  - Fort Myers, Florida
  - Hallandale, Florida
  - Hialeah, Florida
  - Jacksonville, Florida
  - Leesburg, Florida
  - Miami, Florida
  - Orlando, Florida
  - Sunrise, Florida
  - West Palm Beach, Florida
  - Columbus, Georgia
  - Park Ridge, Illinois
  - Wichita, Kansas
  - Baton Rouge, Louisiana
  - Bangor, Maine
  - Newton, Massachusetts
  - Plymouth, Massachusetts
  - Flowood, Mississippi
  - Hattiesburg, Mississippi
  - Creve Coeur, Missouri
  - Princeton, New Jersey
  - Springfield, New Jersey
  - Albuquerque, New Mexico
  - Brooklyn, New York
  - Cedarhurst, New York
  - Latham, New York
  - Staten Island, New York
  - Charlotte, North Carolina
  - Wilmington, North Carolina
  - Oklahoma City, Oklahoma
  - Portland, Oregon
  - Norristown, Pennsylvania
  - Plains, Pennsylvania
  - East Providence, Rhode Island
  - San Antonio, Texas
  - Salt Lake City, Utah
  - Bennington, Vermont
  - Charlottesville, Virginia
  - Williamsburg, Virginia
  - Richland, Washington
- Geelong, Victoria, Australia
- Leuven, Belgium
- Canada (4):
  - Kelowna, British Columbia
  - Halifax, Nova Scotia
  - Chatham, Ontario
  - Toronto, Ontario
- Czechia (2):
  - Prague
  - Rychnov nad Kněžnou
- Milan, Lombardy, Italy
- Amsterdam, Netherlands
- Poland (2):
  - Bialystok
  - Warsaw
- South Africa (6):
  - Johannesburg, Gauteng
  - Pretoria, Gauteng
  - Durban, KwaZulu-Natal
  - Bellville, Western Cape
  - George, Western Cape
  - Somerset West, Western Cape
- South Korea (3):
  - Busan
  - Incheon
  - Seoul
- Spain (4):
  - Terrassa, Barcelona
  - Burgos
  - Madrid
  - Salamanca
- United Kingdom (5):
  - Glasgow
  - Isleworth
  - Northampton
  - Penarth
  - Southampton